CLINICAL TRIAL: NCT04366362
Title: Anterior Cruciate Ligament Surgical Reconstruction Based on Individualized Musculoskeletal Models: a Randomized Control Trial
Brief Title: Individualized Anterior Cruciate Ligament Versus Conventional Reconstruction
Acronym: IACLR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgios Chalatsis, MD, MSc, PhD Cand, Resident in Orthopaedics, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC1
Record Dates: First submitted 2019-06-10; First posted 2020-04-28 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL; Anterior; Cruciate; Ligament; Reconstruction; Individualised; Anatomical; Navigation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Two groups of patients, randomly assigned
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be aware of the group that they will be part of. Assessors before and after surgery will not be aware of patients groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convetional reconstruction group (Active Comparator): Patients will undergo ACL reconstruction based on conventional ACL surgery
  Interventions: Procedure: Conventional ACL reconstruction
- Individualised reconstruction group (Experimental): Patients will undergo ACL reconstruction based on their special anatomical and functional characteristics and with the use of a navigation system
  Interventions: Procedure: Individualised ACL reconstruction

INTERVENTIONS:
Procedure: Individualised ACL reconstruction — ACL reconstruction based on anatomical and functional distinctiveness of each patient separately
  Arms: Individualised reconstruction group
Procedure: Conventional ACL reconstruction — ACL reconstruction based on surgeons experience without taking into account any other patients characteristics
  Arms: Convetional reconstruction group

SUMMARY:
A randomised prospective control trial comparing the efficiency of a more individualized approach in ACL reconstruction with the help of neuromuscular computer models with traditional ACL reconstruction practices.

DETAILED DESCRIPTION:
Until now the ACL reconstruction was based on the surgeon's experience. An individualised ACL reconstruction is customized based on each patient's special characteristics. Preoperative and intraoperative evaluation of the native ACL (both anteromedial and posterolateral bundles), knee anatomy and function, level of activity and generalised ligamentous laxity are assessed. Femoral and tibial tunnels should be placed in their anatomical location accounting for both the native ACL insertion site and bony landmarks. Two groups will be created, one with patients undergoing ACL reconstruction based on a surgeon's experience and one based on a more individualised approach according to the particular characteristics of each patient separately. In addition, patients in the second group will undergo ACL reconstruction with the use of Computer Assisted System (Navigation).

Preoperatively and postoperatively, the patients will be assessed with the KT2000 system, the KOOS (Knee injury and Osteoarthritis Outcome), the Tegner- Lysholm Knee scoring system and the IKDC (International Knee Documentation Committee). Additionally, all patient will be examined for their knee function with the use of a 3D gait analysis system.

The follow-up examination will take place 6 and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACL rupture undergoing ACL reconstruction surgery with closed epiphyses, younger than 45 years old

Exclusion Criteria:

* No previous surgery in the knee (except partial meniscectomy), no major systematic pathology

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of the change of stability of the operated knee between the two groups from Baseline until 1 year post-operation | Baseline and 1 year post operation
  Participants in two groups will be assessed with KT2000 arthrometer before and after ACL reconstruction regarding knee stability. Additionally knee kinematics and gait analysis before and after the ACL reconstruction will be compared between the two groups in a gait analysis lab.

SECONDARY OUTCOMES:
Compare the change from Baseline between the patients of the two groups in KOOS (Knee Injury & Osteoarthritis Outcome) from the baseline until 1 year post operation | Baseline and 1 year post operation
  Originally published in 1998 in The Journal of Orthopaedic and Sports Physical Therapy, the Knee injury and Osteoarthritis Outcome Score (KOOS) assesses patient pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sport and recreation (5 items), and knee related quality of life (4 items). Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms. The KOOS is a patient reported joint-specific score, which may be useful for assessing changes in knee pathology over time, with or without treatment.
Compare the change from Baseline between the patients of the two groups in IKDC (International Knee Documentation Committee Subjective Knee Form) from the baseline until 1 year post operation. | Baseline and 1 year post operation
  the International Knee Documentation Committee Subjective Knee Form (IKDC) was designed to assess patients with a variety of knee disorders including ligamentous and meniscal injuries as well as patellofemoral pain and osteoarthritis. The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Compare the change from Baseline between the patients of the two groups in Tegner Lysholm Knee Scoring Scale from the baseline until 1 year post operation. | Baseline and 1 year post operation
  Lysholm Knee Scoring Scale was designed to be used for evaluating outcomes of knee ligament surgery, particularly for symptoms related to instability. The Lyshom Knee Scoring Scale is a patient-reported instrument that consists of subscales for pain, instability, locking, swelling, limp, stair climbing, squatting, and the need for support. Scores range from 0 (worse disability) to 100 (less disability).
Compare the post operation MRI of the 2 groups | 1 year post operation
  Evaluate tunnel positioning in femur and tibia and the graft integration and compare them between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hantes, MD, Study Chair — University General Hospital of Larissa
Locations (1):
- Michael Hantes, Larissa, Greece